CLINICAL TRIAL: NCT04633772
Title: Randomized Clinical Trial Phase I/II for the Use of Angiotensin-(1-7) in the Treatment of Severe Infection by Sars-CoV-2
Brief Title: Use of Angiotensin-(1-7) in COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: Federal University of Minas Gerais (Other); Angitec (Unknown); Fonds Erasme pour la Recherche Medicale (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RBR-35734p
Record Dates: First submitted 2020-11-06; First posted 2020-11-18 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Infection, Coronavirus; Respiratory Failure
Keywords: angiotensin-(1-7); ARDS; renin angiotensin system
MeSH Terms: conditions — Coronavirus Infections; Respiratory Insufficiency | interventions — angiotensin I (1-7)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Angiotensin-(1-7) (Experimental)
  Interventions: Drug: Angiotensin-(1-7)

INTERVENTIONS:
Drug: Angiotensin-(1-7) — Intravenous supplementation of Angiotensin-(1-7)
  Arms: Angiotensin-(1-7)
Drug: Placebo — NaCl 0.9%
  Arms: Placebo

SUMMARY:
The renin-angiotensin system (RAS) has a relevant role in COVID-19, as the virus will enter host's cells via the angiotensin-converting enzyme 2 (ACE2); RAS disequilibrium might also play a key role in the modulation of the inflammatory response that characterizes the lung involvement. Angiotensin-(1-7) is a peptide that could be altered in COVID-19 patient and its supplementation may potentially helpful in this setting.

DETAILED DESCRIPTION:
A novel Coronavirus (SARS-CoV-2) described in late 2019 in Wuhan, China, has led to a pandemic and to a specific coronavirus-related disease (COVID-19), which is mainly characterized by a respiratory involvement. While researching for a vaccine has been started, effective therapeutic solutions are urgently needed to face this threaten. The renin-angiotensin system (RAS) has a relevant role in COVID-19, as the virus will enter host's cells via the angiotensin-converting enzyme 2 (ACE2); RAS disequilibrium might also play a key role in the modulation of the inflammatory response that characterizes the lung involvement. Angiotensin-(1-7) is a peptide that could be altered in COVID-19 patient and it may potentially improve respiratory function in this setting. This a randomized, controlled, investigator-initiated Phase I/Phase II trial is conceived to test the safety and the efficacy of intravenous angiotensin-(1-7) infusion in COVID-19 patients with severe pneumonia admitted to the intensive care unit (ICU). The first phase of the study, with a limited number of patients (n=30) will serve to confirm the safety of the intravenous infusion of the drug by observing the incidence of the adverse events (phase I, open label). In a second phase of the study, conducted in a double-blind manner and including a larger cohort of patients (n=100, Phase II), patients will be randomly assigned to receive either an Angiotensin-(1-7) infusion or placebo. The primary endpoint of the study will be the number of supplemental oxygen-free days by day 28. Secondary outcomes will include length of hospital stay, ICU and hospital free days, ICU and hospital mortality, need for mechanical ventilation, weaning time from mechanical ventilation if intubated, secondary infections, vasopressor needs, changes in PaO2 / FiO2, incidence of deep vein thrombosis, changes in inflammatory markers, plasma levels of angiotensin II and angiotensin (1-7) and radiological findings.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the Intensive Care Unit with severe pneumonia criteria (clinical signs of pneumonia + one of the following criteria: respiratory rate greater than 30/minute; signs of respiratory effort, SatO2 < 90% in room air);
* COVID-19 confirmed or highly suspicious (positive contact or suggestive image)

Exclusion Criteria:

* Diagnosed with cancer (at any stage);
* Hemodynamic instability (need for vasopressors);
* Pregnant women; Immunocompromised patients;
* Palliative Care;
* Inclusion in any other interventionist study;
* Heart failure as a predominant cause of acute respiratory failure;
* Decompensated liver cirrhosis;
* HIV +;
* Dialysis;
* Home / long-term oxygen therapy;
* Idiopathic pulmonary fibrosis

Ages: 17 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
supplemental oxygen-free days (SOFDs) | 28 days
  28 - x, where x = number of days on which the patient is released from supplemental oxygen therapy after start

SECONDARY OUTCOMES:
Hospital length of stay | through study completion, on average 60 days
  Hospital length of stay
ventilator free days | 28 days
  composite outcome of mortality and necessity of mechanical ventilation
ICU free days | through study completion, on average 40 days
  number of days free from intensive care unit
RAS effectors levels | Baseline, 3 and 24 hours after randomization and 72 hours after randomization
  Ang II and Ang-(1-7) circulating levels using mass spectrometry
CT scan findings | through study completion, on average 30 days
  CT scan evolutions compared to baseline including findings compatible with late pulmonary fibrosis.
Changes in inflammatory markers: C reactive protein | through study completion, on average 30 days
  C-reactive protein levels daily measurements
Changes in clinical state: vasopressors usage | through study completion, on average 30 days
  use of vasopressors during hospitalization
Chest X ray findings | through study completion, on average 30 days
  Chest X-ray modifications until hospital discharge
Changes in inflammatory markers: chemokines | Baseline, 3 and 24 hours after randomization and 72 hours after randomization
  pro-inflammatory chemokine levels (IL-1/IL-6) at baseline day 3 and 7
Changes in inflammatory markers: troponin | Baseline, 3 and 24 hours after randomization and 72 hours after randomization
  Troponin plasmatic levels
Changes in thrombotic markers: D-Dimer | Baseline, 3 and 24 hours after randomization and 72 hours after randomization
  D-Dimer
Changes in clinical state: secondary infections | through study completion, on average 30 days
  Secondary infections recorded during hospitalization
Changes in clinical state: deep venous thrombosis | through study completion, on average 30 days
  deep venous thrombosis recorded during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Robson AS Santos, Principal Investigator — Angitex; Ana Martins Valle, Principal Investigator — Federal University of Minas Gerais; Filippo Annoni, Principal Investigator — Erasme University Hospital
Locations (2):
- Brazil (2):
  - Hospital Eduardo de Menezes, Belo Horizonte, Minas Gerais
  - Hospital Mater Dei, Belo Horizonte, Minas Gerais

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martins ALV, Annoni F, da Silva FA, Bolais-Ramos L, de Oliveira GC, Ribeiro RC, Diniz MML, Silva TGF, Pinheiro BD, Rodrigues NA, Dos Santos Matos AH, Motta-Santos D, Campagnole-Santos MJ, Verano-Braga T, Taccone FS, Santos RAS. Angiotensin-(1-7) infusion in COVID-19 patients admitted to the ICU: a seamless phase 1-2 randomized clinical trial. Ann Intensive Care. 2024 Sep 4;14(1):139. doi: 10.1186/s13613-024-01369-0. PMID 39231898